CLINICAL TRIAL: NCT01039896
Title: An Open-label, Randomized, Crossover Study to Evaluate the Safety and Pharmacokinetics After Multiple Administration of SLM0807 Alone and Multiple Co-administration of HKB0701/SLM0807 in Korean Healthy Subjects
Brief Title: A Drug Interaction Study of SLM0807 and HKB0701 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_VCM_101
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group1 (Experimental): SLM0807
  Interventions: Drug: Period I : SLM0807, Period II : HKB0701 and SLM0807
- Group2 (Experimental): SLM0807 and HKB0701
  Interventions: Drug: Period I : HKB0710 and SLM0807, Period II : SLM0807

INTERVENTIONS:
Drug: Period I : SLM0807, Period II : HKB0701 and SLM0807
  Arms: Group1
Drug: Period I : HKB0710 and SLM0807, Period II : SLM0807
  Arms: Group2

SUMMARY:
The aim of this study is to assess whether HKB0701 alters pharmacokinetics of SLM0807.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who are in age range of 20-50years and the weight range is not exceed ±20% of ideal weight. Ideal weight = [height -100]*0.9
* Subjects with no history of any significant chronic disease
* Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data
* Available for the entire study period
* Willing to adhere to protocol requirements and sign a informed consent form.

Exclusion Criteria:

* Subjects who have taken any drugs to induce or inhibit hepatic enzyme activity within 30days prior to drug administration
* Subjects who have symptom of an acute illness within 4 weeks prior to drug administration
* Subjects with a history of clinically significant allergies including drug allergies
* Subjects whose clinical laboratory test values are outside the accepted normal range(Especially,AST or ALT >1.25 times to normal range or total bilirubin > 1.5times to normal range)
* Subjects with a history of drug, caffeine or alcohol abuse (caffeine drink >5cups /day, alcohol >30g/day)
* Heavy smoker ( >10cigarettes/day)
* Subjects who have had a diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice)
* Subjects who have donated plasma within 60days prior to drug administration
* Subjects who have participated in a clinical study within 90days prior to drug administration
* Subjects who have received any drugs that might confound the results of the trial in the opinion of principal investigator (cimetidine within 7days prior to drug administration)
* Female subjects who are pregnant, breastfeeding or not using medically acceptable birth control

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Css,max and AUCinf | up to 24hrs

SECONDARY OUTCOMES:
AUCtau, AUCt, Tmax | up to 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: Jae Gook Shin, MD, ph D, Principal Investigator — Inje University

REFERENCES:
- [Derived] Kim HS, Oh M, Kim EJ, Song GS, Ghim JL, Shon JH, Kim DH, Shin JG. Effect of voglibose on the pharmacokinetics of metformin in healthy Korean subjects. Int J Clin Pharmacol Ther. 2014 Nov;52(11):1005-11. doi: 10.5414/CP202160. PMID 25161160